CLINICAL TRIAL: NCT03329703
Title: The Feasibility of Project UPLIFT for the Treatment of Psychogenic Non-Epileptic Seizures
Brief Title: Project UPLIFT for Psychogenic Non-Epileptic Seizures
Acronym: PNES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Lindsay M. Schommer, Adv Prac Nrs, Neurology, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D17161
Record Dates: First submitted 2017-10-20; First posted 2017-11-06 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Psychogenic Non-Epileptic Seizure; Depression; Non-Epileptic Seizure; Psychogenic Seizure
Keywords: PNES; UPLIFT; Depression; Mindfulness; CBT; Managing Epilepsy Well (MEW) Network; Psychogenic Seizures; Non-Epileptic Seizures
MeSH Terms: conditions — Psychogenic Nonepileptic Seizures; Depression; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate-Treatment (Experimental): This group will receive Project UPLIFT immediately after completing surveys.
  Interventions: Behavioral: Project UPLIFT
- Waitlist Control (Active Comparator): This group will receive Project UPLIFT after waiting approximately 3 months to begin the intervention.
  Interventions: Behavioral: Project UPLIFT

INTERVENTIONS:
Behavioral: Project UPLIFT — A group, telephone-based intervention for depression that uses techniques from mindfulness-based therapy and cognitive therapy. The intervention consists of 8 sessions occurring at the same time and day every week.

SUMMARY:
Developed by researchers from the Centers for Disease Control and Prevention (CDC), Project UPLIFT (Using Practice and Learning to Increase Favorable Thoughts) is a group telephone program designed to improve depression for people with epilepsy. Project UPLIFT uses evidence-based approaches of cognitive-behavioral therapy (CBT) and mindfulness-based cognitive therapy to help people manage and prevent symptoms of depression.

For people with psychogenic non-epileptic seizures, there are few treatment options for depression that address the relationship between mood and seizures. There is evidence that mindfulness-based therapy and cognitive therapy are both effective for people with non-epileptic seizures, both in treating depression and reducing seizure frequency. In this study, Project UPLIFT will be offered to patients with psychogenic non-epileptic seizures.

Project UPLIFT is facilitated by a trained clinician to groups of 4-8 patients over the telephone. The group will meet at a regular time, once a week, for 8 consecutive weeks. Participants will be assigned to one of two groups: an immediate-treatment or a waitlist control group which will begin Project UPLIFT 3 months after enrolling in the study.

DETAILED DESCRIPTION:
Upon enrollment in the study, participants will be randomly assigned to one of two groups: an immediate-treatment group, or a 3-month waitlist control group. Both groups will be given surveys to complete online, and a seizure calendar to keep track of auras, seizures, and events. The immediate-treatment group will be scheduled to start Project UPLIFT with their trained facilitator. Each of the eight weekly sessions will take place at the same day of the week and at the same time, and will last approximately one hour. Participants will have the option of using a fake-name during the telephone calls to conceal their identity during the group telephone calls.

After the 8 weekly sessions, both groups will be given a second set of online surveys to complete individually. At this time, the waitlist control group will be scheduled to start Project UPLIFT with the trained facilitator. After the waitlist group completes the final session of Project UPLIFT, both groups will complete a third and final set of online surveys, thus concluding all study procedures.

ELIGIBILITY:
Inclusion Criteria:

* History of psychogenic non-epileptic seizures, confirmed by study investigator.
* Literate
* Reliable telephone access

Exclusion Criteria:

* Dual diagnosis of PNES with epilepsy.
* Presence of serious mental illness that will impair ability to participate.
* Presence of active suicidal ideation at baseline with intention to act.
* Severe mental disability or estimated intelligent quotient (IQ) less than 70.
* No reliable telephone access.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-23 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
80% of participants who begin Session 1 of UPLIFT will complete 80% of the sessions. | 6 months
  To test the feasibility of giving Project UPLIFT to patients with PNES

SECONDARY OUTCOMES:
Change in depression (Patient Health Questionnaire-9) before and after intervention. | 6 months
  Change from baseline in depression scores, as reported in the Patient Health Questionnaire-9. The PHQ-9 provides a total depression score ranging from 0-27, with higher score indicating more severe depression symptoms.
Change in seizure frequency as assessed by self-report seizure questionnaire. | 6 months
  Change from baseline in seizure frequency on the self-report seizure questionnaire. The self-report seizure questionnaire asks participants to report the number of seizures they have had in the previous week, month, and year. There is no upper limit of the scale, and is not a standardized survey.
Change in anxiety (Generalized Anxiety Disorder-7) before and after the intervention. | 6 months
  Change from baseline in anxiety scores, as reported on the Generalized Anxiety Disorder -7 survey. The GAD-7 provides a total score ranging from 0-21, with a higher score indicating more severe anxiety symptoms.
Change in symptoms of Post-Traumatic Stress Disorder (PTSD Checklist-Civilian Version, PCL-C) before and after the intervention. | 6 months
  Change from baseline in Post-Traumatic Stress Disorder scores as measured by the Post-Traumatic Stress Disorder Checklist - Civilian Version. The PCL-C provides a total score of PTSD severity that ranges from 17-85, with higher score indicating higher symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Schommer, APRN, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) are not planned to be shared without outside researchers.